CLINICAL TRIAL: NCT02768987
Title: Bright 1 Bodies: Extending the Bright Bodies Weight Management Program to Adolescents With Type 1 Diabetes
Brief Title: Bright 1 Bodies Weight Management Program
Acronym: B1B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of the West of Scotland (Other); Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1605017843
Record Dates: First submitted 2016-05-04; First posted 2016-05-11 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: exercise; physical activity; behavior modification; coping skills; self management; glycemic control; overweight; obesity; body composition; adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overweight (Experimental): Sedentary adolescents with T1D and overweight
  Interventions: Behavioral: Bright 1 Bodies
- Normal Weight (Experimental): Sedentary adolescents with T1D and normal weight
  Interventions: Behavioral: Bright 1 Bodies

INTERVENTIONS:
Behavioral: Bright 1 Bodies — A 12-week intensive lifestyle program utilizing group exercise classes adapted for this population, supplemented with coping skills training and diabetes self-management education.

SUMMARY:
Physical inactivity occurs among 65% to 95% of youth with type 1 diabetes (T1D) and based upon limited evidence may contribute to the rapidly growing incidence of overweight among this population. The purpose of the present study is to pilot test a 12-week intensive lifestyle program for adolescents with overweight and T1D utilizing group exercise classes adapted for this population, supplemented with coping skills training and diabetes self-management education to address problem solving behaviors that limit their physical activity and weight control. Our primary aim is to evaluate the changes in physical activity adherence, anthropometrics, and self-management behaviors following this program among sedentary adolescents with T1D and overweight (n=25, OW) compared with sedentary adolescents with T1D and normal weight (n=25, NW). We hypothesize that the OW group will achieve improve physical activity adherence and anthropometrics to the same or greater extent as the NW group and previous Bright Bodies cohorts, and that these changes will correlate with improved exercise-related problem solving. Our secondary aim is to evaluate changes in adipocytokines and epigenetic factors related to the etiology of overweight/obesity following our physical activity intervention. We hypothesize changes in these biomarkers will correlate with changes in anthropometry variables and partially explain any differences in response between the groups and individuals should those occur.

DETAILED DESCRIPTION:
Prevalence of overweight among patients with type 1 diabetes (T1D) of all ages has grown at alarming rates since the 1980s. Physical inactivity occurs among 65% to 95% of youth with T1D and doubles their risk of overweight. A major factor limiting their physical activity appears to be self-managed problem solving around exercise such as adjustments to insulin and diet, which is practiced regularly by less than half of our adolescent patients with T1D and less frequently than any other self-management behavior. Our previous interventions applying coping skills training (ABCs of Diabetes and TeenCope) as well as diabetes self-management (Managing Diabetes) successfully improved problem-solving and other aspects of self-management along with health outcomes among adolescents with T1D, but did not focus on those who were overweight nor promotion of physical activity and weight loss. The Yale Bright Bodies intensive lifestyle program successfully promotes physical activity and weight loss, enrolling >100 overweight youth from greater New Haven annually but does not presently accommodate those with T1D.

The purpose of the present study is to pilot test a 12-week intensive lifestyle program for adolescents with overweight and T1D utilizing group exercise classes from Bright Bodies adapted for this population, supplemented with coping skills training and diabetes self-management education to address problem solving behaviors that limit their physical activity and weight control. Our primary aim is to evaluate the changes in physical activity adherence, anthropometrics (body mass index percentile for age, body fat percentage), and self-management behaviors following this 12-week lifestyles program among sedentary adolescents with T1D and overweight (n=25, OW) compared with sedentary adolescents with T1D and normal weight (n=25, NW). We hypothesize that the OW group will achieve improve physical activity adherence and anthropometrics to the same or greater extent as the NW group and previous Bright Bodies cohorts, and that these changes will correlate with improved exercise-related problem solving.

Although physical activity is recommended for weight loss, outcomes from increased physical activity have been heterogeneously distributed-not all overweight participants lose weight and some even gain weight. Furthermore the etiologies of overweight/obesity and T1D appear to interact, yet no study has tested the influence of physical activity upon biological pathways related to overweight/obesity for patients with T1D. Accordingly, our secondary aim is to evaluate changes in adipocytokines and epigenetic factors related to the etiology of overweight/obesity following our physical activity intervention. We hypothesize changes in these biomarkers will correlate with changes in anthropometry variables and partially explain any differences in response between the groups and individuals should those occur.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the Yale-New Haven Hospital (YNHH) Pediatrics Long Wharf or Trumbull Diabetes Clinic
* Diagnosed with T1D
* 11 to 19 years old
* Sedentary (exercise less than twice per week over past two months)
* n=25 overweight (BMI > 85th percentile for age and sex according to Centers for Disease Control Growth Charts) and n=25 normal weight
* Family willing to commit the time and effort to a family-based lifestyle program.

Exclusion Criteria:

* Endocrinopathies other than type 1 diabetes; adequately treated hypothyroidism, as demonstrated by normal thyroid tests within previous six months, is allowed.
* Concurrent use of systemic (oral, parenteral) glucocorticoids or other medications known to contribute to obesity; inhaled steroids are allowed.
* Any use of pharmacological intervention for weight management, including prescription medication, over the counter medication, or herbal supplements.
* Chronic disease or physical disability that would influence treatment intervention or preclude participation in regular physical activity (e.g., chronic renal failure).
* Psychological conditions such as uncontrolled eating disorder, psychosis, personality disorders and other disorders that will interfere with the ability to maintain complete follow up and adherence to protocol.
* Any concurrent membership in a comprehensive weight management program.
* Inability or unwillingness of the parent to accompany the child to nutrition classes.
* Pregnancy

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline body mass index (BMI) over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline in daily physical activity energy expenditure over 24 weeks | Baseline, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Change from baseline in Progressive Aerobic Cardiovascular Endurance Run score over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline in blood pressure over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline daily insulin usage over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline lipid profile over 12 weeks | Baseline, 12 weeks
Change from baseline adipocytokines over 12 weeks | Baseline, 12 weeks
Change from baseline inflammatory factors including C-reactive protein, interleukin-6, fibrinogen, and plasminogen activator inhibitor-1 over 12 weeks | Baseline, 12 weeks
Change from baseline micro RNA expression over 12 weeks | Baseline, 12 weeks
Change from baseline pediatric quality of life questionnaire score over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline diabetes self-care inventory score over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline hypoglycemia fear survey score over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline psychosocial determinants of physical activity behavior questionnaire score over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline self-perception profile for adolescents questionnaire social acceptance subscale score over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline in handgrip strength over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline in sit-and-reach test over 24 weeks | Baseline, 12 weeks, 24 weeks
Change from baseline in push-up test over 24 weeks | Baseline, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Garrett I Ash, PhD, CSCS, Principal Investigator — Yale University
Locations (1):
- Yale Children's Diabetes Program, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided